CLINICAL TRIAL: NCT07254455
Title: Catheter Ablation Versus Standard Conventional Treatment in Atrial Fibrillation Patients With Heart Failure With Mildly Reduced and Preserved Left Ventricular Ejection Fraction - A Prospective, Randomized, Multi-national Study Using Two Systems for Rhythm Monitoring
Brief Title: CASTLE-HFpEF (Catheter Ablation for Atrial Fibrillation Patients With Heart Failure With Mildly Reduced and Preserved Ejection Fraction)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Boston Scientific Corporation (Industry); Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26-0025
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation; Heart Failure With Preserved Ejection Fraction
Keywords: A-fib; HFpEF; HFmrEF; AF; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard medical therapy for heart failure with preserved ejection fraction arm (No Intervention): Participants randomized to receive medical treatment will be treated according to locally applicable guidelines for standard of care. The choice of the specific pharmacological treatment will be left to the discretion of the treating physician whether it is a rate or rhythm control based on the clinical picture, but maintenance of sinus rhythm through anti arrhythmic drugs (AADs) in this study arm will be encouraged. Electrical cardioversion using a defibrillator is allowed in this study arm.
  Medical therapy for HFmrEF/HFpEF will be continued following standard of care.
- Catheter ablation arm (Experimental): Participants assigned to CA will undergo the procedure as soon as possible after baseline evaluation (within 5 weeks), following the Heart Rhythm Society (HRS) consensus statement using pulsed field ablation (PFA). The main aim of the procedure is to achieve isolation of all four pulmonary veins (PVs).
  In participants with paroxysmal AF, only pulmonary vein isolation (PVI) will be performed. In participants with persistent AF, posterior wall isolation (PWI) in addition to PVI will be applied.
  Medical therapy for HFmrEF/HFpEF will be continued following standard of care. The physician performing the CA must have performed at least 50 prior AF ablation procedures, comprising PVI and PVI +, with the same approach.
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — A catheter ablation (CA) is a minimally invasive medical procedure for treatment of cardiac arrhythmias. Rhythm control of AF is attempted by pulmonary vein isolation (PVI) and posterior wall isolation (PWI). During the procedure, a catheter is guided to the heart through a blood vessel, which is either the femoral vein or a central vein, in order to ablate abnormal conductive heart tissue that causes the arrhythmias. Ablation is achieved either by thermal (cauterization by radiofrequency (RF) ablation / freezing by cryoballoon) or non-thermal mechanisms (primarily irreversible electroporation (IRE) through pulsed field ablation (PFA)). In case of successful ablation, a normal heart rhythm (sinus rhythm) can be restored.
  Arms: Catheter ablation arm

SUMMARY:
The clinical equipoise in the treatment of Atrial Fibrillation (AF) in patients with Heart Failure with mildly reduced Ejection Fraction/Heart Failure with Preserved Ejection Fraction (HFmrEF/HFpEF) reflects the scarcity of randomized trials on different treatment modalities. By generating high-quality, evidence-based, randomized data on the impact of treatment on hard outcomes, Catheter Ablation Versus Standard Conventional Treatment in Atrial Fibrillation Patients with Heart Failure with Preserved Ejection Fraction (CASTLE-HFpEF) will provide clinical decision-making guidance and help physicians in the management of patients with HFmrEF/HFpEF and AF.

The main hypothesis is that Catheter Ablation (CA) for AF is associated with improved clinical outcomes in patients with HFmrEF/HFpEF and AF compared to medical AF treatment strategies on top of optimal medical HF treatment. CASTLE-HFpEF aims to study these hard clinical outcomes in a randomized cohort of patients with AF and HFmrEF/HFpEF.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is highly prevalent and often coexists with atrial fibrillation (AF), but the optimal management strategy for AF in this population remains unclear. The CASTLE-HFpEF (CASTLE-AF II) trial is a prospective, randomized, multicenter study designed to evaluate whether catheter ablation of AF improves clinical outcomes compared with optimized medical therapy in patients with HFpEF.

Approximately 4,000 patients with HFpEF will undergo AF screening using an insertable cardiac monitor. Of these, 980 patients with newly diagnosed AF or AF detected during screening and with an AF burden > 1% will be randomized 1:1 to catheter ablation or guideline-directed medical therapy. All randomized patients will be followed for three years and monitored continuously for AF burden.

The primary endpoint is a hierarchical composite including all-cause mortality, stroke or transient ischemic attack, hospitalization for worsening heart failure, and a clinically meaningful reduction in N-terminal pro-B-type natriuretic peptide (NT-proBNP) at 12 months. Secondary endpoints include total heart failure events, patient-reported quality-of-life outcomes, AF burden and rhythm control metrics, and echocardiographic measures of cardiac structure and function.

This study seeks to determine whether AF ablation improves clinical outcomes and quality of life in patients with HFpEF and AF, and to define the role of rhythm control strategies in this population.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at screening visit.
2. Clinical signs and symptoms of HF (26).
3. Left ventricular ejection fraction (LVEF) >40% within the past 12 months (most recent LVEF measurement)
4. Elevated NT-proBNP levels during screening or within 12 months prior to screening (most recent value; blood test):

   * For patients in normal sinus rhythm (NSR) at the time of blood sampling: NT proBNP ≥300 pg/mL
   * For patients in AF at the time of blood sampling: NT-proBNP ≥600 pg/mL
5. Echocardiographic evidence of HFmrEF/HFpEF, with at least one of the following during screening or within the 12 months prior to screening:

   1. Left atrial volume index (LAVI) ≥34 mL/m2 for patients in NSR, or LAVI ≥40 mL/m2 for patients in AF.
   2. Tricuspid regurgitation (TR) peak velocity >2.8 m/s.
   3. Mitral E/e' ratio at rest ≥9.
   4. Left ventricular mass index (LVMI) ≥115 g/m2 for men and ≥95 g/m2 for women.
   5. Septal thickness or posterior wall thickness ≥1.1 cm.
6. Patients previously diagnosed with persistent AF since ≤4 months prior to screening with an indication for anticoagulation, OR Patients previously diagnosed with paroxysmal AF since ≤4 months prior to screening with an already known AF burden of ≥1% and/or an AF episode of ≥24 hours, with an indication for anticoagulation OR Patients with paroxysmal AF without known AF burden (diagnosed since ≤4 months prior to screening) or no previously diagnosed AF who are subsequently diagnosed with AF after receiving a single-lead electrocardiography (ECG) patch for 30 days. These patients should have an AF burden of ≥1% and/or an AF episode of ≥24 hours on the ECG patch (more details down below in section 8.1.1) and an indication for anticoagulation.
7. Stable optimal medical therapy for HFmrEF/HFpEF for at least 4 weeks (diuretics & SGLT2 inhibitors unless contraindicated; angiotensin receptor-neprilysin inhibitors & mineralocorticoid receptor antagonists as deemed appropriate by the treating physician; Amiodarone and Beta-blockers are not considered for defining heart failure therapy).
8. Signed written informed consent obtained from the participant or participant's legal representative and ability for participant to comply with the requirements of the study.

Exclusion Criteria:

* Participants will be excluded from the study for any of the following reasons:

  1. Previous catheter ablation for AF.
  2. Known infiltrative cardiomyopathy, hypertrophic cardiomyopathy and amyloidosis.
  3. Documented left atrial diameter >6cm.
  4. Any contraindication for chronic anticoagulation therapy or heparin, including hypersensitivity to any of the components.
  5. Acute coronary syndrome, cardiac surgery, angioplasty, or cerebrovascular accident within 2 months prior to enrollment.
  6. Planned cardiovascular intervention during the follow-up period.
  7. Patients with severe valvular disease
  8. Life expectancy ≤12 months.
  9. Untreated hypothyroidism or hyperthyroidism (blood test).
  10. Requirement for dialysis due to end-stage chronic kidney disease.
  11. Mental or physical inability to participate in the study.
  12. Women currently pregnant (blood test) or breastfeeding or not using reliable contraceptive measures during fertility age.
  13. Enrollment in another investigational drug or device study within the last 30 days before registration.
  14. Medical or psychological conditions that would not permit the participant to complete the study or sign informed consent.
  15. Known alcohol or drug abuse.
  16. Presence of a condition, abnormality or disease that in the opinion of the investigator would compromise the safety of the participant or the quality of the data.
  17. Legal incapacity or limited legal capacity.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of all-cause mortality, stroke or transient ischemic attack (TIA), and hospitalizations for worsening HF and clinically relevant decrease of NT proBNP (after 12 months) | Baseline, 12 Months, 36 months
  Hierarchical composite endpoint of the hard outcomes all-cause mortality, stroke or TIA, and hospitalizations for worsening HF (all after 36 months), and clinically relevant decrease of NT proBNP (after 12 months), analyzed using the Win Ratio method for each AF treatment arm (PFA-based CA versus conventional therapy). The Win Ratio is a statistical method designed to analyze composite outcomes with hierarchical clinical priorities, such as death, hospitalization, and functional status.
  Each patient in the treatment group is then compared to each patient in the control group, forming all possible unmatched pairs. Within each pair, the patient who experiences the more favorable outcome at the highest priority level is declared the "winner." The Win Ratio is calculated as the total number of wins in the treatment group divided by the number of wins in the control group, providing a clinically intuitive summary of net benefit.

SECONDARY OUTCOMES:
Combined hard outcomes (all-cause mortality, stroke or TIA, hospitalizations for worsening HF; time to first event) | 36 months
  The combined hard outcome is defined as the time to the first occurrence of any of the three specified components, and will be analyzed using Kaplan-Meier survival curves and the log-rank test to compare event-free survival between groups.
Total HF-related events (hospitalization for worsening HF and outpatient worsening HF events) | 36 months
  The investigators will count the total HF-related events (hospitalization for worsening HF and outpatient worsening HF events) until the end of study. It will be tested via Poisson regression or negative binomial regression, according to the data distribution. Which model to use will be determined from the likelihood ratio test.
  To analyze how often the HF-related events happen. Depending on how the data looks, the investigators will choose between two models - one called Poisson regression and the other called negative binomial regression. To decide which model fits the data better, the investigators will use a statistical method called a "likelihood ratio test," which compares the two models and tells the investigators which one works best for the data.
Kansas City Cardiomyopathy Questionnaire (KCCQ) score | Baseline, 3 Months, 6 months, 12 months, 24 months, 36 months
  Kansas City Cardiomyopathy Questionnaire (KCCQ) score will be tested by t-test or the Wilcoxon test, according to normal distribution or not determined by the Wil-Shapiro test. KCCQ is a validated, patient-reported outcome measure designed to assess health status in individuals with heart failure. It evaluates multiple domains, including physical limitation, symptom frequency and severity, social function, self-efficacy, and quality of life. Scores range from 0 to 100, with higher scores indicating better health status. The KCCQ is sensitive to clinical changes and is widely used in both clinical trials and practice to measure the impact of heart failure treatments from the patient's perspective. A change of 5-10 points is generally considered clinically meaningful.
All-cause mortality (time to event) | 36 Months
  All-cause mortality will be tested via Kaplan-Meier curve and Log-rank test. The investigators will measure the survival rate based on the time to event.
Stroke or TIA (time to event) | 36 Months
  Stroke or TIA (time to event): tested via Kaplan-Meier curve and Log-rank test. The investigators will measure the first event a stroke or TIA has happened based on the time to event.

CONTACTS AND LOCATIONS:
Overall Officials: Nassir Marrouche, MD, Principal Investigator — Tulane University

IPD SHARING:
Plan to Share IPD: No